CLINICAL TRIAL: NCT02648893
Title: Effect Of Delivering Micronutrients Through Multiple Biofortified Food Crops On Nutritional Status And Immune Function: A Feeding Trial In The First 1000 Days Of Life In India
Brief Title: Effect Of Multiple Biofortified Food Crops On Micronutrient Status And Immune Function Among Indian Infants and Their Mothers
Acronym: MBFC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cornell University (Other)
Collaborators: SNDT Women's University (Other); Arogyavaram Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB #: 1508005782
Record Dates: First submitted 2015-11-23; First posted 2016-01-07 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Vitamin A Deficiency; Iron Deficiency; Zinc Deficiency
Keywords: iron; zinc; vitamin A; biofortified; efficacy; India; infant; trial
MeSH Terms: conditions — Vitamin A Deficiency; Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBFC-Exp (Experimental): The MBFC-Exp (Multiple biofortified food crops - Experimental) arm will consume meals based on biofortified food crops.
  Interventions: Other: Multiple biofortified food crops (MBFC-Exp)
- MBFC-C (Active Comparator): The MBFC-C (Multiple biofortified food crops - Control) arm will consume the same meals based on non-biofortified (commercially available) food crops.
  Interventions: Other: Commercially available non-fortified food crops (MBFC-C)

INTERVENTIONS:
Other: Multiple biofortified food crops (MBFC-Exp) — Meals from three biofortified food crops will be consumed by children (and potentially their lactating mothers) three times per day, six days per week, for 9 months.
  Other Names: Biofortified food crops
  Arms: MBFC-Exp
Other: Commercially available non-fortified food crops (MBFC-C) — This arm will consume meals based on three commercially available (non-biofortified) food crops three times per day, six days per week, for 9 months.
  Other Names: Non-biofortified food crops
  Arms: MBFC-C

SUMMARY:
In this study, meals based on multiple food crops (containing either biofortified or commercially-available food crops) will be fed to young children in Madanapalle, Andhra Pradesh, India over a period of nine months to measure growth, cognitive changes, and immune function in comparison to children receiving non-biofortified crops. Mothers of the participating children will also be included in the study.

DETAILED DESCRIPTION:
Iron, zinc, and vitamin A deficiency remain a major worldwide public health problem especially in developing countries such as India. In this randomized study, 200 children aged 6-12 months (and their lactating mothers) from Madanapalle, Andhra Pradesh, India will be fed meals based on (either biofortified or commercially-available) multiple food crops three times per day, six days per week, for nine months. We will recruit children from 6 - 24 months of age. The goal of this study is to examine the effects of the biofortified multiple food crops on immune function, growth, and cognitive function in this age group. The key outcome measures are biomarkers of vitamin A, iron and zinc status, growth (anthropometric z-scores), and immune and cognitive function. Nutrient biomarkers will be assessed at enrollment (baseline), at an intermediate time point (midline; random serial sampling) and after 9 months of follow-up (endline). Additionally, we will measure concentrations of C-reactive protein (CRP) and alpha 1-acid glycoprotein (AGP), as iron and zinc biomarkers can be influenced by inflammation. To assess cognitive function, multiple specific aspects of memory and attention will be assessed. Higher-level, integrative cognitive abilities that require the coordination of multiple specific functions, such as problem-solving and exploratory behavior and global aspects of attention during free play with toys, will also be assessed. In addition, the Development Assessment Scales for Indian Infants (DASII) test will be conducted at baseline, intermediate, and endline assessments to obtain a broad measure of attainment of developmental milestones that can be used to compare the characteristics of this cohort with those reported in the literature.

ELIGIBILITY:
Inclusion Criteria

Children: Age 6 to 24 months (at enrollment);

Mothers: Biological mothers of included children.

Exclusion Criteria

Children

* Age below 6 months or above 24 months (at time of screening);
* Hemoglobin <9 g/dL (at time of screening);
* Presence of severe malnutrition according to Wellcome Classification (marasmus, marasmic kwashiorkor, kwashiorkor, weight-for-height z-score < -3);
* Prior known or current diagnoses of HIV/AIDS, Malaria, Dengue fever, Tuberculosis;
* Children whose biological mother is unable to bring her/him to feeding center daily;
* Possibility of migrating out of the study catchment area for more than 4 consecutive weeks;
* Prior or current consumption of iron, zinc, and/or vitamin A supplements;
* Any known dietary allergies.

Mothers

- Severe anemia (Hemoglobin <7g/ dL)

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2019-02-28 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Biomarkers of vitamin A, iron, and zinc status | endline (9 months)
  Determined by serum ferritin (ng/mL) after nine months' intervention.
Biomarkers of vitamin A, iron, and zinc status | endline (9 months)
  Determined by sTfR (soluble Transferrin Receptor; mg/L) after nine months' intervention.
Biomarkers of vitamin A, iron, and zinc status | endline (9 months)
  Determined by serum retinol (µmol/L) after nine months' intervention.
Biomarkers of vitamin A, iron, and zinc status | endline (9 months)
  Determined by serum zinc (mcg/mL) after nine months' intervention.
Biomarkers of vitamin A, iron, and zinc status | endline (9 months)
  Determined by RBP (Retinol-binding Protein; ng/mL) after nine months' intervention.
Biomarkers of vitamin A, iron, and zinc status | endline (9 months)
  Determined by hemoglobin (g/dL) after nine months' intervention.
Biomarkers of vitamin A, iron, and zinc status | endline (9 months)
  Determined by hepcidin (ng/mL) after nine months' intervention.
Biomarkers of vitamin A, iron, and zinc status | endline (9 months)
  Determined by CRP (mg/L) after nine months' intervention.
Biomarkers of vitamin A, iron, and zinc status | endline (9 months)
  Determined by AGP (mg/L) after nine months' intervention.
Physical growth | endline (9 months)
  As determined by length/height (cm) after nine months' intervention.
Physical growth | endline (9 months)
  As determined by weight (kg) after nine months' intervention.
Physical growth | endline (9 months)
  As determined by head circumference (cm) after nine months' intervention.
Physical growth | endline (9 months)
  As determined by mid-upper arm circumference (mm) after nine months' intervention.
Immune function | endline (9 months)
  As assessed by cytokines and vaccine response after 9 months of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh Mehta, MBBS, ScD, Principal Investigator — Cornell University; Julia L. Finkelstein, ScD, Principal Investigator — Cornell University; Shobha Udipi, PhD, Principal Investigator — SNDT Women's University; Bonam Wesley, MBBS, Principal Investigator — Arogyavaram Medical Centre; Jere D Haas, PhD, Principal Investigator — Cornell University
Locations (2):
- India (2):
  - Arogyavaram Medical Centre, Madanapalle
  - S.N.D.T. Women's University, Mumbai

IPD SHARING:
Plan to Share IPD: No